CLINICAL TRIAL: NCT06562361
Title: A First-In-Human, Microdosing, Clinical Trial to Investigate Binding of the PET Tracer [68Ga]Ga-DOTA-CYS-ATH001 Targeting PDGFRβ in Healthy Subjects as Compared to Patients With MASH, PSC and CD
Brief Title: A Microdose Trial Investigating Binding of [68Ga]Ga-DOTA-CYS-ATH001 in Healthy Subjects and Different Patient Groups.
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Antaros Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: INT008; 2023-506555-15-00 (EU CTIS Number)
Record Dates: First submitted 2024-08-14; First posted 2024-08-20 (Actual); Last update posted 2024-08-29 (Actual); Status verified 2024-08

CONDITIONS: MASH; PSC; Fibrostenotic Crohn's Disease; Healthy Volunteers
Keywords: PET; Tracer; PDGFRB; MASH; PSC; MRI; Crohn´s Disease
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 100 µg [68Ga]Ga-DOTA-Cys-ATH001 (target dose of 200 MBq) (Experimental): All participants will receive a single, bolus iv injection of up to 100 µg [68Ga]Ga-DOTA-Cys-ATH001 (target dose of 200 MBq). At Visit 4, cohort 1b (healthy participants, n=3) and cohort 2b (presumed MASH participants, n=3) will come for a second PET/MR imaging visit within 6 weeks from the first imaging visit where an additional bolus iv injection of up to 100 µg [68Ga]Ga-DOTA-Cys-ATH001 will be administered.
  Interventions: Drug: [68Ga]Ga-DOTA-Cys-ATH001

INTERVENTIONS:
Drug: [68Ga]Ga-DOTA-Cys-ATH001 — Target dose of 200MBq [68Ga]Ga-DOTA-Cys-ATH001 corresponding to a maximum mass dose of 100 µg, administered as an intravenous bolus dose.

SUMMARY:
The goal of this clinical trial is to use positron emission tomography (PET) to evaluate and compare the binding of the novel tracer [68Ga]Ga-DOTA-Cys-ATH001 in the liver and/or gastrointestinal tract between healthy volunteers and different patient groups including patients with metabolically caused steatohepatitis (MASH), patients with fibrostenotic Crohn´s Disease (CD) and patients with primary sclerosing cholangitis (PSC).The study will also assess the safety of a microdose of 68Ga]Ga-DOTA-Cys-ATH001 and how it is distributed in different parts of the body. The main questions the study aims to answer are:

* What does the uptake of the [68Ga]Ga-DOTA-Cys-ATH001 PET-tracer look like in the liver of healthy subjects, and in that of patients with MASH and PSC?
* What does the uptake of the [68Ga]Ga-DOTA-Cys-ATH001 PET-tracer look like in the GI tract of healthy subjects, and that of patients with fibrostenotic CD?
* How much [68Ga]Ga-DOTA-Cys-ATH001 PET-tracer can be found in the blood after injection?
* How is [68Ga]Ga-DOTA-Cys-ATH001 uptake distributed in the body?
* What medical problems do participants have when receiving [68Ga]Ga-DOTA-Cys-ATH001?

Participants will:

Receive one administration of [68Ga]Ga-DOTA-Cys-ATH001, after which examination with PET is performed. Magnetic Resonance Imaging (MRI) is also used in the study to create a detailed picture of the body and its function which will facilitate the interpretation of the results of the PET examination. A subset of participants will have blood samples collected after the tracer administration to assess the blood levels of the tracer over time.

A subset of participants will come back for a second visit where they will receive a second administration of [68Ga]Ga-DOTA-Cys-ATH001, followed by PET and MRI.

A health check-up is performed before dosing, and a safety assessment will be performed after dosing. A remote follow-up visit is performed the day after the dosing visit.

DETAILED DESCRIPTION:
This is a first-in-human (FIH), phase 0, multi-center, non-randomized trial to investigate [68Ga]Ga-DOTA-Cys-ATH001 PET-tracer binding in the liver and in the GI tract in healthy subjects and patients with metabolically caused steatohepatitis (MASH), patients with fibrostenotic Crohn´s Disease (CD) and patients with primary sclerosing cholangitis (PSC), in a total of 5 different cohorts, including a sub-trial to assess test-retest reliability and a sub-trial to assess dosimetry. The allocation of cohorts is:

* Cohort 1a (n=3): Healthy volunteers, sub-group dosimetry,
* Cohort 1b (n=3): Healthy volunteers, sub-group test/retest,
* Cohort 2a (n=3): Presumed MASH patients, sub-group dosimetry,
* Cohort 2b (n=3): Presumed MASH patients, sub-group test/retest,
* Cohort 3 (n=6): Verified MASH patients,
* Cohort 4 (n=6): Fibrostenotic CD patients,
* Cohort 5 (n=6): PSC patients.

The participants will come for 2 or 3 visits to the trial site. The screening (Visit 1) will include an eligibility check and review of health status. Participants in cohort 2 and cohort 3 will perform a FibroScan® investigation.

At Visit 2, participants will come to the trial site for PET/MRI and safety assessments. The participants will receive a single, bolus iv injection of a maximum of 100 µg [68Ga]Ga-DOTA-Cys-ATH001 after which participants will be examined by whole-body PET/MRI scans. A sub-group of participants in cohort 1 (cohort 1a, healthy subjects, n=3, the first 3 participants in this cohort) and cohort 2 (cohort 2a, presumed MASH patients, n=3, the first 3 participants in this cohort) will be participating in a sub-trial to calculate the whole-body dosimetry of the tracer. These participants will have one longer PET visit and will be examined by sequential whole-body PET/MRI scans to determine tracer biodistribution and clearance. At Visit 4 (within 6 weeks of Visit 2), participants taking part in the test/retest sub-trial (Cohorts 1b and 2b) will come for a second PET/MRI visit which includes a second administration of [68Ga]Ga-DOTA-Cys-ATH001.

To determine tracer clearance from blood, venous (1a and b and 2a and b) and arterial (1b and 2b) PK samples will be collected post-dose. No PK samples will be taken from cohorts 3 to 5.

Safety assessments will take place after the PET/MRI (vital signs, 12-lead ECG, safety laboratory sampling and injection site reactions). A remote follow-up by telephone (Visit 3) will be performed the day after [68Ga]Ga-DOTA-Cys-ATH001 dosing to follow-up on AEs, injection site reactions and concomitant medication.For participants in cohorts 1b and 2b (the test/retest sub-group), a remote follow-up by telephone (Visit 5) will be performed the day after [68Ga]Ga-DOTA-Cys-ATH001 dosing to follow-up on AEs, injection site reactions and concomitant medication.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to give written informed consent for participation in the trial and able to comply with all trial procedures and requirements.
2. Male or female participant aged 18 to 75 years, inclusive, at the screening visit.
3. Body mass index (BMI) ≥ 19 and < 40.0 kg/m2 at the time of the screening visit.
4. Women of childbearing potential (WOCBP) must practice abstinence from heterosexual intercourse (only allowed when this is the preferred and usual lifestyle of the participant) or must agree to use a highly effective method of contraception with a failure rate of < 1 % to prevent pregnancy from at least 2 weeks prior to administration of tracer for at least 1 week after the PET imaging examination (or for at least 1 weak after the last PET imaging examination for those participants undergoing test/retest PET imaging). In addition, any male partner of a female participant must, unless he has undergone vasectomy, agree to use a condom during the same time period.

   The following are considered highly effective methods of contraception:
   * combined (estrogen and progestogen-containing) hormonal contraception associated with inhibition of ovulation (oral, intravaginal, transdermal),
   * progestogen-only hormonal contraception associated with inhibition of ovulation (oral, injectable, implantable),
   * intra-uterine device [IUD]or intra-uterine hormone-releasing system [IUS]) WOCBP must refrain from donating eggs until 3 months after the last tracer administration.

   WOCBP with an exclusive male partner who has undergone vasectomy may choose not to use contraceptives.

   Women of non-childbearing potential are pre-menopausal females who have undergone any of the following surgical procedures; hysterectomy, bilateral salpingectomy, or bilateral oophorectomy, or who are post-menopausal defined as 12 months of amenorrhea (in questionable cases a blood sample with detection of follicle-stimulating hormone [FSH] >25 IU/L is confirmatory).

   Male participants must be willing to use condom or be vasectomized or practice sexual abstinence from heterosexual intercourse (only allowed when this is the preferred and usual lifestyle of the participant) to prevent pregnancy and drug exposure of a partner and refrain from donating sperm from the administration of tracer until 3 months after the administration of tracer. Any female partner of a non-vasectomized male participant who is of childbearing potential must use contraceptive methods with a failure rate of < 1% to prevent pregnancy (see above) from at least 2 weeks prior to administration of tracer to 4 weeks after administration of tracer.

   Cohort-specific inclusion criteria:

   Cohort 1 (healthy participants)
5. Medically healthy participant without abnormal clinically significant medical history, physical findings, vital signs, ECG, and laboratory values at the time of the screening visit, as judged by the Investigator.

   Cohort 2 (presumed MASH patients) MASH diagnosis based on non-invasive assessments. Participants should have a high level of disease activity with regards to pro-peptide of type III collagen (ProC3) as a marker of ongoing fibrogenesis.
6. Steatosis according to biopsy, radiology, or controlled attenuation parameter (CAP) (≥ 280 dB/M 8), assessments ≤ 24 weeks prior to the screening visit.
7. At least 1 cardiometabolic criteria from the following list:

   A. BMI ≥ 25 kg/m2 [23 Asia] OR waist circumference (WC) > 94 cm (M) 80 cm (F) OR ethnicity adjusted, B. Fasting serum glucose ≥ 5.6 mmol/L [100 mg/dL] OR 2-hour post-load glucose levels ≥ 7.8 mmol/L [≥ 140 mg/dL] OR HbA1c ≥ 5.7% [39 mmol/L) OR type 2 diabetes OR treatment for type 2 diabetes, C. Blood pressure ≥ 130/85 mmHg OR specific antihypertensive drug treatment, D. Plasma triglycerides ≥ 1.70 mmol/L [150 mg/dL] OR lipid-lowering treatment, E. Plasma high-density lipoprotein (HDL)-cholesterol ≤ 1.0 mmol/L [40 mg/dL] (M) and ≤ 1.3 mmol/L [50 mg/dL] (F) OR lipid-lowering treatment.
8. ProC3 ≥ 12.6 ng/mL. Cohort 3 (verified MASH patients) MASH diagnosis based on historical liver biopsy. Participants should have a high level of disease activity with regards to ProC3 as a marker of ongoing fibrogenesis, to allow for correlation to PET-tracer uptake.
9. Evidence of steatosis according to biopsy, radiology, or CAP (≥ 280 dB/M) or MRI-PDFF, assessments ≤ 24 weeks prior to the screening visit.
10. At least 1 cardiometabolic criteria from the following list:

    A. BMI ≥ 25 kg/m2 [23 Asia] OR WC > 94 cm (M) 80 cm (F) OR ethnicity adjusted, B. Fasting serum glucose ≥ 5.6 mmol/L [100 mg/dL] OR 2-hour post-load glucose levels ≥ 7.8 mmol/L [≥ 140 mg/dL] OR HbA1c ≥ 5.7% [39 mmol/L) OR type 2 diabetes OR treatment for type 2 diabetes, C. Blood pressure ≥ 130/85 mmHg OR specific antihypertensive drug treatment, D. Plasma triglycerides ≥ 1.70 mmol/L [150 mg/dL] lipid-lowering treatment, E. Plasma HDL-cholesterol ≤ 1.0 mmol/L [40 mg/dL] (M) and ≤ 1.3 mmol/L [50 mg/dL] (F) OR lipid-lowering treatment.
11. Historical liver biopsy 24 weeks to 4 weeks prior to inclusion with histologically proven metabolic dysfunction-associated steatotic liver disease (MASLD).
12. ProC3 ≥ 12.6 ng/mL. Cohort 4 (fibrostenotic CD patients)
13. Fibrostenotic CD as evidenced by persistent luminal narrowing with or without obstructive symptoms as assessed with MRI, ≤ 24 weeks prior to the screening visit OR fibrostenotic CD by positive colonoscopy up to 24 weeks prior to the screening visit.
14. Crohn's disease activity index (CDAI) < 150
15. Calprotectin < 250
16. C-reactive protein (CRP) < 20 Cohort 5 (PSC patients)
17. Large duct PSC, including intrahepatic bile duct involvement, according to MRI/MRCP.
18. ProC3 ≥ 12.6 ng/mL

Exclusion Criteria:

1. Any contraindication for MRI according to a standard checklist used in clinical practice, including claustrophobia, metallic implants or internal electrical devices (e.g., cochlear implant, nerve stimulator, gastric pacemaker, bladder stimulator, cardiac pacemaker, defibrillator, artificial valves in heart, aneurysm clips or coils, etc.), inability to stay in supine position for 90 minutes, and permanent makeup or tattoos which in the Investigator's opinion might jeopardize the participant's safety or interfere with the imaging assessments.
2. Having worked as a metal worker or welder.
3. History of any clinically significant disease or disorder which, in the opinion of the Investigator, may either put the participant at risk because of participation in the trial or influence the results or the participant's ability to participate in the trial.
4. Any clinically significant illness, medical/surgical procedure, or trauma within 4 weeks of the screening visit.
5. Any malignancy within the past 12 months before the screening visit, with the exception of successfully treated basal cell carcinoma of the skin or in situ prostate cancer under active surveillance, with no interventions scheduled during the period of trial participation.
6. Any planned major surgery within the duration of the trial participation.
7. Participants who are pregnant, currently breastfeeding, or intend to become pregnant during the course of the trial.
8. Any positive result at the screening visit for serum hepatitis B surface antigen, hepatitis B or C antibodies and/or human immunodeficiency virus (HIV).
9. Any chronic active infection (e.g., HIV, Hepatitis B or C, tuberculosis, etc.).
10. Poor peripheral venous access, as judged by the Investigator.
11. After 10 minutes of supine rest at the screening visit, any vital signs values outside the following ranges:

    * Systolic blood pressure: < 90 or >165 mmHg, or
    * Diastolic blood pressure < 50 or >100 mmHg, or
    * Pulse < 40 or > 90 bpm
12. The participant has a change in body weight ≥5%, 3 months before the screening visit.
13. The participant has any laboratory abnormality or condition that, in the Investigator's opinion, could adversely affect the safety of the participant or impair the assessment of trial results.
14. Clinically significantly abnormal 12-lead ECG recording result or cardiac symptoms as judged by the Investigator.
15. The participant is using any prohibited concomitant medications as described in the protocol, at the discretion of the Investigator.
16. Current use of any hormone therapy at doses that may cause metabolic interference as judged by the Investigator. Stable hormonal replacement therapy is allowed.
17. Currently participating, or previous participation in another clinical trial within 30 days prior to the screening visit or previous participation in another PET imaging trial within the last 12 months.
18. Positive screening result for alcohol at the screening visit (cohorts 1a and 1b only).
19. Ongoing or previous alcohol abuse, or long-standing excessive intake of alcohol, as judged by the Investigator.
20. Presence or history of drug abuse, as judged by the Investigator.
21. History of, or current use of anabolic steroids, as judged by the Investigator.
22. Plasma donation within 1 month of screening or blood donation (or corresponding blood loss) during the last 3 months prior to screening.
23. The Investigator considers the participant unlikely to comply with trial procedures, restrictions, and requirements.

    Additional exclusion criteria for all participants (cohorts 2-5):
24. The participant is receiving treatment with vitamin E, thiazolidinediones, or glucagon-like peptide-1 receptor agonists unless on a stable dose for 3 months before the screening Visit and is anticipated to maintain the same dosing regimen throughout trial participation.
25. Participants with HbA1c ≥48 mmol/mol (6.5%) at screening without a previous diagnosis of T2D must not take part in the study. Participants with a previous diagnosis of T2D are permitted to enter the study if on a stable regimen of antidiabetic therapy for at least 3 months before screening. Participants who are on a stable regimen of antidiabetic therapy for at least 3 months before screening and have HbA1c of ≥ 63 mmol/mol (9%) at screening should be excluded.
26. Clinically significant disease, apart from T2D, which in the opinion of the Investigator might interfere with the interpretation of the trial results and/or the safety of the participant, or in any other way unsuitable for participation in this clinical trial.
27. The participant has a severe immune-mediated inflammatory disease (IMID) (e.g., rheumatoid arthritis, spondylarthritis disease spectrum, connective tissue disorders, cutaneous inflammatory conditions such as psoriasis, atopic dermatitis, hidradenitis suppurativa, asthma, multiple sclerosis). Participants with inactive IMID or active IMID of mild to moderate severity are permitted to enter the trial.

    Additional exclusion criteria for MASH and PSC participants (cohorts 2-3, and 5)
28. Liver stiffness > 25 kPa by transient elastography or any sign of decompensation. For cohorts 2 and 3, based on the FibroScan® evaluation on the screening visit, and for cohort 5 based on routine elastography performed ≤ 12 months.
29. For participants with biopsy-confirmed fibrosis stage F2 or F3, the participant has any of the following during the screening period:

    * Aspartate aminotransferase (AST) levels > 5 x the upper limit of normal (ULN).
    * Alanine aminotransferase (ALT) levels > 5 x ULN.
    * Alkaline phosphatase (ALP) ≥ 2 x ULN (cohorts 2 and 3) and ALP ≥ 10 (cohort 5).
    * Serum creatinine ≥1.5 x ULN or has an estimated glomerular filtration rate (eGFR) < 45 mL/min/1.73m2 (the revised Lund-Malmö GFR estimating equation will be used).
    * International normalized ratio (INR) >1.3.
    * Total TBL ≥ULN (except for patients with a documented history of Gilbert's syndrome if direct bilirubin is within the normal reference range).
    * Direct bilirubin ≥ 3 x ULN.
    * Platelet count < 60 x 109/L.
    * Presence or history of ascites, hepatic encephalopathy, or variceal bleeding.
    * Presence or history of Child-Pugh > 6 (Class B or C), unless due to therapeutic anticoagulation.
    * Presence or history of Model for End-Stage Liver disease (MELD) score >12 (only for cohorts 2-3).

    Note: It is the Investigator's decision, in consultation with the Sponsor, to allow participants to enter the study who have clinically meaningful rising tendencies in liver chemistries or significantly elevated liver chemistries that do not yet satisfy but could be interpreted as clinically concerning (i.e., AST or ALT > 4 x ULN) at any visit during the screening period.
30. The participant has a change in body weight ≥ 5% after qualifying liver biopsy. Additional criteria for fibrostenotic CD participants (cohort 4)
31. MRI findings consistent with only inflammation, i.e., edema, hyperemic intestinal wall, restricted diffusion, mesenteric lymphadenopathy etc.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-08 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
[68Ga]Ga-DOTA-Cys-ATH001 uptake in the whole liver of healthy subjects compared with patients with MASH and PSC | Assessed during the intervention
  Difference in [68Ga]Ga-DOTA-Cys-ATH001 mean standardized uptake value (SUV) in the whole liver of healthy subjects (cohort 1), compared with patients with MASH (cohort 2 and 3) and PSC patients (cohort 5).
[68Ga]Ga-DOTA-Cys-ATH001 uptake in the GI tract of healthy subjects compared with patients with fibrostenotic CD | Assessed during the intervention
  Difference in [68Ga]Ga-DOTA-Cys-ATH001 SUV in the GI tract of healthy subjects (cohort 1) compared with patients with fibrostenotic CD (cohort 4).

SECONDARY OUTCOMES:
[68Ga]Ga-DOTA-Cys-ATH001 PET-tracer PK in arterial and venous plasma | Assessed 5 minutes to 125 minutes post-dose
  [68Ga]Ga-DOTA-Cys-ATH001 PET-tracer PK (radioactivity associated with the parent compound) in arterial and venous plasma for up to 125 minutes after injection.

OTHER OUTCOMES:
Whole-body dosimetry of [68Ga]Ga-DOTA-Cys-ATH001 PET tracer in healthy subjects and patients with presumed MASH. | Assessed during the intervention
  Whole-body dosimetry of [68Ga]Ga-DOTA-Cys-ATH001 PET tracer in healthy subjects (cohort 1a) and patients with presumed MASH (cohort 2a).
Safety of [68Ga]Ga-DOTA-Cys-ATH001 PET tracer | Assessed up to 48 hours post intervention
  Safety of [68Ga]Ga-DOTA-Cys-ATH001 PET tracer as assessed by
  * Frequency of, seriousness, and intensity of AEs.
  * Frequency of clinically significant changes in vital signs, ECG, safety laboratory measurements (hematology, clinical chemistry, coagulation, and urinalysis) and physical examination findings.
  * Frequency of injection site reactions.

CONTACTS AND LOCATIONS:
Overall Officials: Johan Vessby, Principal Investigator — Section of Gastroenterology/Hepatology SE-751 85 Uppsala, Sweden
Locations (3):
- Sweden (3):
  - CTC Karolinska, Stockholm
  - CTC Akademiska Uppsala University Hospital, Entrance 85, 2nd level, Uppsala
  - Section of Gastroenterology/Hepatology, Uppsala University Hospital, Uppsala

IPD SHARING:
Plan to Share IPD: No